CLINICAL TRIAL: NCT00351702
Title: Evaluation of Two Different Preventive Therapy Regimens for Tuberculosis in HIV Infected Persons
Brief Title: Preventive Therapy for Tuberculosis in HIV Infected Persons
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr C Padmapriyadarsini, Director, Tuberculosis Research Centre, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: trc20B
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Human Immunodeficiency Virus; Tuberculosis
Keywords: Preventive therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis | interventions — Isoniazid; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isoniazid (Active Comparator): Isoniazid (300mg) daily for 36 months
  Interventions: Drug: Isoniazid with Ethambutol
- Isoniazid + Ethambutol (Experimental): Isoniazid (300 mg) + Ethambutol (800 mg) daily for 6 months
  Interventions: Drug: Isoniazid with Ethambutol

INTERVENTIONS:
Drug: Isoniazid with Ethambutol — Isoniazid (300mg) with Ethambutol (800mg) daily for 6 months

SUMMARY:
Title: Evaluation of efficacy of two different preventive therapy regimens for tuberculosis in HIV infected persons

Phase: Phase III trial

Population: 650 HIV positive patients without tuberculosis

Number of sites: Three

1. Tuberculosis Research centre, Chennai
2. Government General Hospital, Chennai
3. Government Rajaji Hospital, Madurai

Study Duration: 36 months

Study Objectives: To compare the efficacy of two TB preventive therapy regimens in reducing the incidence of tuberculosis and mortality among HIV-infected persons

Study Design:

The study will be a two-armed prospective randomized clinical trial among HIV- positive patients without active tuberculosis. Enrolled patients will be assigned to one of the two unsupervised self-administered treatment regimens i.e. EH for 6 months or INH alone for 3 years. At the end of a 3-year follow-up, incidence of TB and overall mortality will be compared in each group.

Study Endpoints:The primary end point of the study will be development of tuberculosis and the secondary endpoints will include adverse drug reactions and mortality rate.

DETAILED DESCRIPTION:
Study population and enrollment:

All HIV positive patients seeking care at one of the study centers, above the age of 15 years, not suffering from a serious illness, non-pregnant, and in whom TB was ruled out using the enhanced screening process, will be enrolled in the study. The consent form for prophylaxis trial will be read to the patients in the local language and written consent will be obtained from willing patients

Randomization and Dosing:

All patients enrolled in the prevention trial will be randomized to one of the study groups using a permuted block randomization scheme of four. Stratification will be done by Mantoux reading (>5mm and ≤5mm). The group assignment list will be generated centrally before the start of trial and sequentially numbered sealed envelopes containing the study group assigned will be prepared independently. At the initiation of prophylaxis, each patient will be counseled about the importance of taking drugs regularly. Patients will be asked to return the empty packets as well as unused tablets at each monthly visit.

The treatment regimens in each study group will be as follows:

1. Ethambutol (800 mg) and Isoniazid (300 mg) daily for six months, self-administered, collected once in fifteen days.
2. Isoniazid (300 mg) daily for 3 years with fortnightly collection of drugs Subjects in both study groups will receive 10 mg of Pyridoxine daily during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 15 years
2. HIV positivity (on 2 different ELISA tests on the same blood sample)
3. Living in Chennai or Madurai within a defined area of intake - 25 km radius.
4. Likely to remain in the same area for at least three years after start of treatment
5. The patient is judged to be cooperative and willing for fortnightly attendance for the next 3 years
6. Is agreeable for home visits
7. No major complications of HIV disease like encephalopathy, renal or hepatic disease or end stage disease.
8. No other medical condition that might interfere with management like diabetes, convulsions, serious cardiac disease.
9. Patients who fulfill laboratory criteria (hemoglobin > 7.0g/l,granulocyte count>11,000/l, platelet count > 1 lakh/l. serum alanine amino transferase concentration < 2.5 times the upper limit of normal and serum creatinine concentration < 1.1 mgs%, random blood sugar < 140 mgs%) will be enrolled into the study.

Exclusion Criteria:

1. Resides outside area of intake.
2. Pregnancy and lactation.
3. Patients with major psychiatric illnesses and severe depression
4. Major complications of HIV disease like encephalopathy, renal or hepatic disease or end stage disease
5. Serious cardiac disease (CCF, IHD), uncontrolled diabetes mellitus, convulsions, cancer, moribund state
6. Previous antituberculosis treatment for more than 1 month
7. Patients on ART -

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 683 (Actual)
Dates: Start 2001-02; Primary Completion 2008-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure is the development of tuberculosis. | September 2008

SECONDARY OUTCOMES:
Secondary outcome measures include adverse drug reactions and mortality rate. | September 2008

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Swaminathan, MD MNAMS, Principal Investigator — Tuberculosis Research Centre, India
Locations (1):
- Tuberculosis Research Centre, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Bucher HC, Griffith LE, Guyatt GH, Sudre P, Naef M, Sendi P, Battegay M. Isoniazid prophylaxis for tuberculosis in HIV infection: a meta-analysis of randomized controlled trials. AIDS. 1999 Mar 11;13(4):501-7. doi: 10.1097/00002030-199903110-00009. PMID 10197379
- [Background] Wilkinson D, Squire SB, Garner P. Effect of preventive treatment for tuberculosis in adults infected with HIV: systematic review of randomised placebo controlled trials. BMJ. 1998 Sep 5;317(7159):625-9. doi: 10.1136/bmj.317.7159.625. PMID 9727988
- [Background] Hawken MP, Meme HK, Elliott LC, Chakaya JM, Morris JS, Githui WA, Juma ES, Odhiambo JA, Thiong'o LN, Kimari JN, Ngugi EN, Bwayo JJ, Gilks CF, Plummer FA, Porter JD, Nunn PP, McAdam KP. Isoniazid preventive therapy for tuberculosis in HIV-1-infected adults: results of a randomized controlled trial. AIDS. 1997 Jun;11(7):875-82. doi: 10.1097/00002030-199707000-00006. PMID 9189212
- [Background] Whalen CC, Johnson JL, Okwera A, Hom DL, Huebner R, Mugyenyi P, Mugerwa RD, Ellner JJ. A trial of three regimens to prevent tuberculosis in Ugandan adults infected with the human immunodeficiency virus. Uganda-Case Western Reserve University Research Collaboration. N Engl J Med. 1997 Sep 18;337(12):801-8. doi: 10.1056/NEJM199709183371201. PMID 9295239
- [Background] Gordin F, Chaisson RE, Matts JP, Miller C, de Lourdes Garcia M, Hafner R, Valdespino JL, Coberly J, Schechter M, Klukowicz AJ, Barry MA, O'Brien RJ. Rifampin and pyrazinamide vs isoniazid for prevention of tuberculosis in HIV-infected persons: an international randomized trial. Terry Beirn Community Programs for Clinical Research on AIDS, the Adult AIDS Clinical Trials Group, the Pan American Health Organization, and the Centers for Disease Control and Prevention Study Group. JAMA. 2000 Mar 15;283(11):1445-50. doi: 10.1001/jama.283.11.1445. PMID 10732934
- [Result] Swaminathan S, Menon PA, Gopalan N, Perumal V, Santhanakrishnan RK, Ramachandran R, Chinnaiyan P, Iliayas S, Chandrasekaran P, Navaneethapandian PD, Elangovan T, Pho MT, Wares F, Paranji Ramaiyengar N. Efficacy of a six-month versus a 36-month regimen for prevention of tuberculosis in HIV-infected persons in India: a randomized clinical trial. PLoS One. 2012;7(12):e47400. doi: 10.1371/journal.pone.0047400. Epub 2012 Dec 14. PMID 23251327
- Available data/document: published manuscript — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0047400 — the study has been published and has been provided in the citation. the paper conatins the required information regarding study results and conclusion